CLINICAL TRIAL: NCT04830137
Title: A Phase 1, Dose Escalation, Safety and Tolerability Study of NX-2127, a Bruton's Tyrosine Kinase (BTK) Degrader, in Adults With Relapsed/Refractory B-cell Malignancies
Brief Title: A Study of NX-2127 in Adults With Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NX-2127-001
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Waldenstrom Macroglobulinemia (WM); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); Follicular Lymphoma (FL); Diffuse Large B-cell Lymphoma (DLBCL); Primary Central Nervous System Lymphoma (PCNSL)
Keywords: BTK Degrader; BTK Inhibitor; B-cell Malignancy; Lymphoma; IMiD; Lenalidomide; Pomalidomide; Bruton's Tyrosine Kinase; NX-2127; Targeted Protein Degradation; Chimeric Targeting Molecule (CTM); C481; C481S
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Phase 1a Dose Escalation (Experimental): Multiple dose levels of NX-2127 to be evaluated; determination of MTD/Phase 1b recommended dose
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 1 in CLL or SLL (Dose A) (Experimental): CLL/SLL patients whose disease has failed treatment with a BTK inhibitor
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 1 in MCL (Dose A) (Experimental): MCL patients whose disease has failed treatment with a BTK inhibitor and an anti-CD20 monoclonal antibody (mAb) based regimen
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 1 in FL, MZL or WM (Dose A) (Experimental): FL or MZL patients whose disease has failed treatment with an anti-CD20 mAb-based regimen; or WM whose disease has failed treatment with a BTK inhibitor
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 1 in DLBCL (Dose A) (Experimental): DLBCL patients whose disease has failed treatment with an anti-CD20 mAb-based regimen and either: an anthracycline-based regimen; or an anti-CD19-based regimen; or another/palliative regimen
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 1 in PCNSL (Dose A) (Experimental): PCNSL patients whose disease has failed at least 1 prior line of treatment
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 2 in CLL or SLL (Randomized to Dose A or Dose B) (Experimental): CLL/SLL patients whose disease has failed treatment with a BTK inhibitor
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 2 in MCL (Randomized to Dose A or Dose B) (Experimental): MCL patients whose disease has failed treatment with a BTK inhibitor and an anti-CD20 monoclonal antibody (mAb) based regimen
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 2 in FL, MZL or WM (Randomized to Dose A or Dose B) (Experimental): FL or MZL patients whose disease has failed treatment with an anti-CD20 mAb-based regimen; or WM whose disease has failed treatment with a BTK inhibitor
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 2 in DLBCL (Randomized to Dose A or Dose B) (Experimental): DLBCL patients whose disease has failed treatment with an anti-CD20 mAb-based regimen and either: an anthracycline-based regimen; or an anti-CD19-based regimen; or another/palliative regimen
  Interventions: Drug: NX-2127
- Phase 1b Dose Optimization Stage 2 in PCNSL (Randomized to Dose A or Dose B) (Experimental): PCNSL patients whose disease has failed at least 1 prior line of treatment
  Interventions: Drug: NX-2127

INTERVENTIONS:
Drug: NX-2127 — Oral NX-2127

SUMMARY:
This is a first-in-human Phase 1a/1b multicenter, open-label oncology study designed to evaluate the safety and anti-cancer activity of NX-2127 in patients with advanced B-cell malignancies.

DETAILED DESCRIPTION:
Phase 1a (Dose Escalation) will evaluate the safety and tolerability of NX-2127 in adult patients with relapsed/refractory (R/R) B-cell malignancies, who have required and received at least 2 prior systemic therapies (or at least 1 prior therapy for patients with WM or PCNSL) and for which no other therapies are known to provide clinical benefit.

Phase 1b (Dose Optimization) will use a 2-stage design to further investigate the safety, tolerability, and preliminary efficacy of NX-2127 in R/R B-cell malignancies based on the dosage(s) selected in Phase 1a.

Stage 1 will enroll approximately 10 participants per group based on B-cell lymphoma/leukemia indication at a specific dose selected from the first part of the study. The Sponsor may decide to open Stage 2 for any given group after review of safety and anti-tumor activity data from Stage 1.

In Stage 2, an additional 10 participants will be enrolled at the dose from Stage 1 as well as 20 additional participants at a second alternative dose. Participants will be randomly assigned to one of the 2 dose levels in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Patients must have measurable disease per disease-specific response criteria
* Patients with indolent forms of NHL must meet the criteria requiring systemic treatment (i.e., iwCLL, IWG, Lugano Classification of Lymphoma response criteria, or International PCNSL Collaborative Group response criteria)
* Patients with transformed lymphoma are eligible for the study with the exception of those detailed in Exclusion Criteria #1: Prolymphocytic leukemia, MCL with blastoid histology, MCL with pleomorphic morphology, or MCL with known TP53 mutation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (non-PCNSL indications) or 0 - 2 (PCNSL patients)
* Adequate organ and bone marrow function
* Patients of child-bearing potential must use adequate contraceptive measures to avoid pregnancy for the duration of the study as defined in the protocol

Inclusion Criteria for Patients in Phase 1a:

* Have histologically confirmed R/R CLL, SLL, WM, MCL, and MZL, FL, DLBCL, or PCNSL
* Received at least 2 prior systemic therapies (or at least 1 prior therapy for patients with WM or PCNSL) and have no other therapies known to provide clinical benefit
* Must require systemic therapy

Inclusion Criteria for Patients in Phase 1b:

* Must have one of the following histologically documented R/R B-cell malignancies:

  * CLL/SLL whose disease has failed treatment with a BTKi;
  * MCL whose disease has failed treatment with BTKi and an anti-CD20 mAb-based regimen
  * FL or MZL whose disease has failed treatment with an anti-CD20 mAb-based regimen; or WM whose disease has failed treatment with a BTKi
  * PCNSL whose disease failed at least 1 prior line of treatment
  * DLBCL whose disease has failed treatment with an anti-CD20 mAb-based regimen and either: an anthracycline-based regimen; or an anti-CD19-based regimen, or another/ palliative regimen (either progressed post stem cell transplant or transplant-ineligible)

Exclusion Criteria:

* Active, uncontrolled autoimmune hemolytic anemia or autoimmune thrombocytopenia
* History of known/suspected other autoimmune disease (exception(s): patients with alopecia, vitiligo, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at screening are allowed.)
* Unable to swallow capsules or have a condition that may interfere in the delivery, absorption, or metabolism of the study drug
* Bleeding diathesis, or other known risk for acute blood loss
* Patients requiring ongoing treatment with warfarin or an equivalent vitamin K antagonist and within 7 days prior to the first dose of study drug
* Prior radiotherapy within 2 weeks of planned start of study drug (excluding limited palliative radiation)
* Toxicities from previous anticancer therapies must have resolved to baseline levels or to Grade 1 (except for alopecia, hypothyroidism with adequate replacement therapy, hypopituitarism with adequate replacement therapy, peripheral neuropathy or hematologic parameters meeting inclusion criteria).
* Active known second malignancy. Exception: patients with non-metastatic, non-melanoma skin cancer are eligible
* Patient has had major surgery (e.g. requiring general anesthesia) within 4 weeks before the planned first dose of study drug
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2. Exception: patients with well-controlled HIV (e.g., CD4 > 350/mm3 and undetectable viral load) are eligible.
* Current active liver disease from any cause
* Active viral reactivation (e.g., CMV or EBV)
* Use of systemic corticosteroids exceeding 20 mg/day prednisone (or equivalent) for non-PCNSL indications within 15 days prior to the planned start of study drug. PCNSL patients may not exceed corticosteroid doses of 40 mg/day prednisone (or equivalent) and should be on a stable or decreasing dose for 7 days prior to planned study start.
* Use of non-steroidal immunosuppressive drugs within 30 days prior to start of the study
* Clinically significant, uncontrolled cardiac, cardiovascular disease, or history of myocardial infarction within 6 months of planned start of study drug
* Administration of any strong cytochrome P450 3A (CYP3A) inducers or inhibitors for 14 days prior to the first dose of study drug, and any P-glycoprotein inhibitors (for 2 days) or moderate inducers of CYP3A for 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Protocol Specified Dose-Limiting Toxicities | Up to 24 months
  Phase 1a
To establish the MTD and/or recommended Phase 1b dosage(s) of NX-2127 | Up to 24 months
  Phase 1a
To evaluate the clinical activity of NX-2127 at the recommended Phase 1b dosage(s) based on overall response rate (ORR) as assessed by the Investigator | Up to 4 years
  Phase 1b
Number of Participants with Adverse Events and Clinical Laboratory Abnormalities | Up to 5 years
  Phase 1a/1b

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Profile of NX-2127: Maximum Serum Concentration | Up to 5 years
  Phase 1a/1b - Sampling following the first dose, pre and post-dose at selected cycles, and at the end of treatment
Duration of response (DOR) as assessed by the Investigator | Up to 5 years
  Phase 1a/1b
Progression-free survival (PFS) as assessed by the Investigator | Up to 5 years
  Phase 1a/1b
Overall survival (OS) as assessed by the Investigator | Up to 4 years
  Phase 1b
To further evaluate the safety and tolerability of NX-2127 by collecting adverse events, treatment emergent adverse events, and incidence of all deaths | Up to 4 years
  Phase 1b
Complete response (CR) rate / CR with incomplete marrow recovery as assessed by the Investigator | Up to 5 years
  Phase 1a/1b

CONTACTS AND LOCATIONS:
Overall Officials: Paula O'Connor, MD, Study Director — Nurix Therapeutics, Inc.
Locations (16):
- United States (16):
  - City of Hope, Duarte, California
  - University of California Irvine, Orange, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Sarah Cannon Research Institute at Colorado Blood Cancer Institute, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Sarasota, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang D, Harris HM, Chen J, Judy J, James G, Kelly A, McIntosh J, Tenn-McClellan A, Ambing E, Tan YS, Lu H, Gajewski S, Clifton MC, Yung S, Robbins DW, Pirooznia M, Skanland SS, Gaglione E, Mhibik M, Underbayev C, Ahn IE, Sun C, Herman SEM, Noviski M, Wiestner A. NRX-0492 degrades wild-type and C481 mutant BTK and demonstrates in vivo activity in CLL patient-derived xenografts. Blood. 2023 Mar 30;141(13):1584-1596. doi: 10.1182/blood.2022016934. PMID 36375120